CLINICAL TRIAL: NCT02472080
Title: Open Labeled Phase II Study Evaluating Efficacy and Safety of Chemotherapy With Gemcitabine - Oxaliplatin Combination for Advanced Refractory Thyroid Cancer Patients
Brief Title: Gemcitabine - Oxaliplatin for Advanced Refractory Thyroid Cancer Patients: a Phase II Study
Acronym: THYGEMOX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inefficiency
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P130933
Record Dates: First submitted 2015-05-12; First posted 2015-06-15 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2018-03

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine -oxaliplatine combination (Experimental)
  Interventions: Drug: gemcitabine -oxaliplatine combination

INTERVENTIONS:
Drug: gemcitabine -oxaliplatine combination — gemcitabine (2g/50mL)-oxaliplatine (200mg /40mL) combination, IV,every 2 weeks for 8cycles

SUMMARY:
Radioiodine refractory differentiated thyroid cancer is a rare tumor and therapeutic options are limited in this setting. Molecular targeted therapies have recently been developed for progressive disease and demonstrated clinical activity, especially with anti-angiogenic agents.

For patients with contra-indication to these agents or in case of progression or toxicity during treatment, chemotherapy is usually proposed but this strategy has not been validated by prospective data.

The investigators propose to conduct an open single arm phase 2 study to evaluate response rate according to RECIST 1.1 with GEMOX regimen (gemcitabine - oxaliplatin combination) for advanced radioiodine refractory differentiated thyroid cancer patients after anti-angiogenic agents or in case of contra-indication to anti-angiogenic therapy.

DETAILED DESCRIPTION:
The aim is to study efficacy of chemotherapy with gemcitabine - oxaliplatin combination for advanced radioiodine refractory differentiated thyroid cancer patients after anti-angiogenic agents or in case of contra-indication to anti-angiogenic therapy.

For refractory thyroid cancer patients, in case of contra-indication to molecular targeted therapies or in case of progression or toxicity during treatment, alternative treatments are urgently needed.

Our study could precise if cytotoxic agents should remain a treatment option for refractory thyroid cancer after molecular targeted therapies or in case of contra-indication.

Numerous clinical trials are proposed to evaluate various molecular targeted therapies for refractory thyroid cancer, either conducted by institutional or industrial promoters. In contrast, chemotherapy trials are lacking. As generics are actually available for gemcitabine and oxaliplatin, no industrial support can be expected and prospective evaluation a chemotherapy regimen need to be conducted by an institutional promoter ("Assistance Publique - Hôpitaux de Paris"), supported by many French expert teams through the rare tumor network ""TUTHYREF"".

GEMOX regimen will be administrated intravenously every two weeks in ambulatory setting.

The objective of this study is to analyse the efficacy of chemotherapy with gemcitabine - oxaliplatin combination for advanced radioiodine refractory differentiated thyroid cancer patients after anti-angiogenic agents or in case of contra-indication to anti-angiogenic therapy.

The primary end point is overall response rate (complete + partial response - CR+PR), according to RECIST 1.1, assessed by local investigator at 4 months.

30 patients will be included in a two steps design (Fleming design). A response rate lower than 15% define the inefficacy level. Minimal efficacy should be 35% response rate.

First step: inclusion of 15 patients. If 2 or less responses are observed: end of study for inefficacy If 6 or more responses are observed: efficacy endpoint has been reached If 3 to 5 responses are observed, additional inclusions are needed. Second step: inclusion of 15 additional patients. Nine responses are expected to define a positive study. Details are presented in statistical section.

The secondary end points are:

* Safety report according to NCI CTCAE v 4.0 grading scale
* Early metabolic response rate on 18F-FDG-PET/CT at 2 months
* Disease control rate (DCR = CR + PR + SD) ≥ 6 months
* Duration of response
* Time to progression
* Progression free survival
* Overall survival.
* Evolution of quality of life according to Fact-G and EQ-5D "

ELIGIBILITY:
"Main Inclusion criteria

1. Histologically confirmed differentiated or poorly differentiated thyroid cancer that is metastatic or unresectable
2. Patients refractory to radio iodine
3. Radiologic evidence of clinically relevant disease progression (as per RECIST 1.1)
4. Measurable disease (by RECIST Version 1.1 criteria)
5. ECOG performance status of ≤ 1
6. Adequate hematologic, renal and liver function
7. Negative serum pregnancy test in premenopausal women.
8. Signed informed consent

Main Non-Inclusion criteria

1. Other histological subtypes of thyroid tumors: anaplastic, medullary, lymphoma or sarcoma
2. Active CNS metastases
3. Prior chemotherapy. Patients treated previously with molecular targeted therapies could be included.
4. Severe, acute or chronic medical or psychiatric condition or laboratory abnormality which in the judgment of the investigator would make the patient inappropriate for entry into this study"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
overall response rate | 4 months
  overall response rate measured (complete and partial responses) by CT-scan according to RECIST criteria v1.1

SECONDARY OUTCOMES:
number of adverse events and serious adverse events (AE) according to CTCAE v4.03 | up to 12 month
  recording number of adverse events and serious adverse events (AE) according to CTCAE v4.03, during chemotherapy and follow up.
Early metabolic response rate on 18F-FDG-TEP/CT | 2 months
  semi-quantitative PET Response Criteria in Solid Tumors PERCIST1.0 "modified" using SUVmax and body-weight. Central reviewing of FDG-PET data by two readers at the end of the study will be done.
Disease control rate | 4 months
  Disease control rate (DCR) is defined as the percentage of patients who have achieved complete response (CR), partial response (PR) or stable disease (SD).
Time to progression | up to 36 months
  Time from documentation of tumor response to disease progression or date of death from any cause
Progression free survival | up to 36 months
  Time from documentation of tumor response to disease progression or date of death from any cause
Overall survival | up to 36 months
  Delay between inclusion and death from any cause
Quality of life | at day 1(week 1, i.e first cycle) and repeated every 28 days (i.e at W5, W9, W13, W17) during chemotherapy and every 3 months until 12 months
  evolution of quality of life will be assessed by the scores at the FACT-G and EQ-5D surveys (French version)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Leenhardt, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpetriere, Paris, France